CLINICAL TRIAL: NCT01233518
Title: Determination of Fractional Flow Reserve by Anatomic Computed Tomographic Angiography
Acronym: DeFACTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HeartFlow, Inc. (Industry)
Collaborators: Baim Institute for Clinical Research (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-901-001
Record Dates: First submitted 2010-10-13; First posted 2010-11-03 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease
Keywords: CCTA Coronary Artery Disease CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Other): Patients will receive cCTA, ICA, FFR, and cFFR per protocol.
  Interventions: Device: FFR

INTERVENTIONS:
Device: FFR — Fractional flow reserve measured during cardiac catheterization

SUMMARY:
This is a prospective, multi-center trial conducted at up to 20 US, Canadian, European and Asian centers designed to determine the diagnostic performance of CT-FLOW (the investigational technology) by coronary computed tomographic angiography (CCTA) for non-invasive assessment of the hemodynamic significance of coronary lesions, as compared to direct measurement of fractional flow reserve (FFR) during cardiac catheterization as a reference standard.

DETAILED DESCRIPTION:
285 patient, prospective, multi-center trial conducted at up to 20 US, Canadian, European and Asian centers designed to determine the diagnostic performance of CT-FLOW (the investigational technology) by coronary computed tomographic angiography (CCTA) for non-invasive assessment of the hemodynamic significance of coronary lesions, as compared to direct measurement of fractional flow reserve (FFR) during cardiac catheterization as a reference standard

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients providing written informed consent
* Scheduled to undergo clinically-indicated non-emergent invasive coronary angiography (ICA)
* Has undergone >64 multidetector row CCTA within 60 days prior to ICA
* No cardiac interventional therapy between the CCTA and ICA

Exclusion Criteria:

* Prior coronary artery bypass graft (CABG) surgery
* Prior percutaneous coronary intervention (PCI) for which suspected coronary artery lesion(s) are within a stented coronary vessel
* Contraindication to adenosine, including 2nd or 3rd degree heart block; sick sinus syndrome; long QT syndrome; severe hypotension, severe asthma, , severe COPD or bronchodilator-dependent COPD
* Suspicion of acute coronary syndrome (acute myocardial infarction and unstable angina)
* Recent prior myocardial infarction within 40 days of ICA
* Known complex congenital heart disease
* Prior pacemaker or internal defibrillator lead implantation
* Prosthetic heart valve
* Significant arrhythmia or tachycardia
* Impaired chronic renal function (serum creatinine >1.5 mg/dl
* Patients with known anaphylactic allergy to iodinated contrast
* Pregnancy or unknown pregnancy status
* Body mass index >35
* Patient requires an emergent procedure
* Evidence of ongoing or active clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, and severe congestive heart failure (NYHA III or IV) or acute pulmonary edema
* Any active, serious, life-threatening disease with a life expectancy of less than 2 months
* Inability to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James K Min, MD, FACC, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Spring Hill Hospital, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Min JK, Berman DS, Budoff MJ, Jaffer FA, Leipsic J, Leon MB, Mancini GB, Mauri L, Schwartz RS, Shaw LJ. Rationale and design of the DeFACTO (Determination of Fractional Flow Reserve by Anatomic Computed Tomographic AngiOgraphy) study. J Cardiovasc Comput Tomogr. 2011 Sep-Oct;5(5):301-9. doi: 10.1016/j.jcct.2011.08.003. Epub 2011 Aug 7. PMID 21930103
- [Result] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562
- [Derived] Park HB, Heo R, O Hartaigh B, Cho I, Gransar H, Nakazato R, Leipsic J, Mancini GBJ, Koo BK, Otake H, Budoff MJ, Berman DS, Erglis A, Chang HJ, Min JK. Atherosclerotic plaque characteristics by CT angiography identify coronary lesions that cause ischemia: a direct comparison to fractional flow reserve. JACC Cardiovasc Imaging. 2015 Jan;8(1):1-10. doi: 10.1016/j.jcmg.2014.11.002. PMID 25592691

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm Study
Started | 285
Completed | 252
Not Completed | 33

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study
Number analyzed (Participants) | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 135
  >=65 years | 117
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 178
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 92
  Belgium | 43
  Canada | 1
  Latvia | 41
  South Korea | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Diagnostic Accuracy of CCTA Plus FFRCT and CCTA Alone
Description: Diagnostic accuracy of CCTA (Cardiac Computed Tomography Angiography) plus FFRCT (Noninvasive Fractional Flow Reserve computed from CCTA) to determine presence or absence of at least one hemodynamically (HD)-significant coronary artery stenosis* at the subject level using binary outcomes when compared to invasive FFR (Fractional Flow Reserve) as the reference standard. In the per-patient analysis, vessels with the most adverse clinical status were selected to represent a given patient. FFR and FFRCT measurements were recorded on a continuous scale and dichotomized at the 0.80 threshold (values ≤0.80 considered diseased; values >0.80 nondiagnostic for ischemia). Stenosis on CCTA was recorded at the 50% threshold (stenoses ≥50% considered obstructive and <50% as non-significant). Prespecified primary endpoint was expected to be greater than 70% of the lower bound of the 95% confidence interval.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Single Arm Study: Per-patient performance (diagnostic accuracy) CCTA plus FFRCT
Arm/Group | Single Arm Study
Number analyzed (Participants) | 252
percentage of participants
  Accuracy of FFRCT | 73 [67 to 78]
  Accuracy of CCTA | 64 [58 to 70]

2. Secondary Outcome: Diagnostic Performance of CCTA Plus FFRCT at the Subject Level
Description: Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of CCTA plus CT-FLOW at the subject level using binary outcomes when compared to FFR as the reference standard.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 252
percentage of participants
  Sensitivity | 90 [84 to 95]
  Specificity | 54 [46 to 83]
  Positive predictive value | 67 [60 to 74]
  Negative predictive value | 84 [74 to 90]

ADVERSE EVENTS:
Arm/Group | Single Arm Study
Serious Adverse Events (participants affected / at risk) | 2/252
Other Adverse Events (participants affected / at risk) | 0/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=252)
Retroperitoneal bleed (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Septic shock (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No